CLINICAL TRIAL: NCT03646708
Title: Triangular Phenotyping and Response Assessment in Small Bowel Crohn's Disease Using Magnetic Resonance Enterography (MRE) and Novel Proteomic Biomarkers
Brief Title: Response Assessment in SB CD
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Other Study IDs: 201805058
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Small Bowel Crohn's Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SBCD patients starting a new biologic therapy: As part of your standard clinical care (soc), patient will be started on a biologic (anti-tumor necrosis factor (TNF)s, vedolizumab and ustekinumab) based on your interactions with your treating gastroenterologist after standard of care clinical assessment.

SUMMARY:
The small bowel (SB) is involved in ~70% of patients with Crohn's disease (CD). There is an unmet need for accurate and clinically meaningful methods to measure small bowel Crohn's Disease (SBCD) activity. This is particularly relevant as the field moves towards "treat-to-target" management strategies. The overall objective of this proposal is to establish that radiologic transmural response (TR) and a novel proteomic biomarker are accurate and clinically meaningful predictors of SBCD inflammatory activity and response to biologic therapy. To address this objective, we will establish a prospectively followed cohort of SBCD patients starting a new biologic therapy. These patients will be comprehensively phenotyped using state of the art MRE imaging, proteomic profiling and clinical disease activity indices. We will use this innovative approach of triangular phenotyping to address our central hypothesis that "Corticosteroid-free remission at 52 weeks after biologic therapy initiation is predicted by short term radiologic TR or early changes in serum proteomic biomarker profiles". Serum proteomic biomarker profiles will be evaluated using SOMAscanTM (SomaLogic, Inc., Boulder, Colorado, USA), a novel platform allowing high-throughput analysis of proteins through Slow Off-rate Modified DNA Aptamer (SOMAmer)-based capture array. Our preliminary data using SOMAscan identified a panel of 12 serum proteins whose differential expression pattern from Week 0 to week 6 after starting a biologic can predict week 14 clinical remission in SBCD patients. The significance of this proposal is that the development of an early predictive model using radiological and serum endpoints will facilitate a personalized algorithmic approach to identify patients with SBCD who will benefit from treatment escalation or change to a different biologic. Furthermore, it will be used to generate a tangible career tool of a prospectively enrolled patient cohort to further study radiologic and biomarker predictors of response in SBCD. This award will also enhance the career of the principal investigator by facilitating acquisition of an enhanced skill set in clinical research, bioinformatics and biomarker discovery.

DETAILED DESCRIPTION:
Patients entering the study will be evaluated by the investigator for all inclusion and exclusion criteria. Once inclusion and exclusion criteria have been determined, all subjects will sign an Internal Review Board (IRB)/Independent Ethics Committee (IEC) approved consent document, which complies with regulatory requirements, prior to any study activities. Subjects will be given adequate time to read and consider the consent document and all study information. They will have the opportunity to ask questions of the investigator(s) and the study team about the study, as well as risks and benefits, prior to signing the document.

Baseline Visit

Baseline assessments will be collected from the clinical care record from the standard of care visit(s) done most prior to the subject receiving their first dose of biologic All assessments will be done/collected prior to the subject's first does of biologic. The baseline visit will consist of the following:

* Demographic information: Date of birth, gender, and race will be collected.
* Clinical assessment: These assessments will be done by the study team prior to the subject receiving the first dose of vedolizumab.
* Physical Exam Findings: Physical exam findings will be taken from the patient's clinical care record from the standard of care visit most recently preceding the initial dose of vedolizumab. If this data is not available from the visit, the information will be obtained from the subject during a separate visit to the clinic by the study team, and prior to the first dose of vedolizumab.
* Blood Tests (C-reactive, Albumin, Hematocrit, SOMAscan panel
* Stool Collection: At the time of consent, participants will be provided a stool collection kit and asked to collect a small amount of stool when they have a bowel movement, prior to their first dose of biologic, for genetic, microbiome, or biomarker analysis. If the patient is unable to provide a stool sample, permission may be asked to obtain a rectal swab, or a sample collection kit will be mailed to them and asked to mail the stool sample back to us in a prepaid envelope. If the patient is in the hospital and tests have been ordered on their stool, stool may be collected from what is left over after the tests have been completed. The stool will be assigned a unique specimen code. The messenger ribonucleic acid (mRNA) in the stool would be extracted and the genetic expression profile of this sample would be determined. All participants consent to having details from their medical records (age, ethnicity, medications, surgery, tobacco use, family history, disease activity, disease history) at the Washington University Medical Center (WUSM), and entered into a database associated with a patient code. If the patient's records do not include all relevant information, a study team member may obtain this information directly from the patient.

The specimen(s) will not have the participant name or address on it; it will be labeled with a code in order to protect the patient's health information and identity. The specimen(s) will be stored in locked freezers in a locked laboratory at WUSM. All coded specimens will be linked to study participants on a separate master list, which will be stored in a locked cabinet (the study coordinators have the only key) or a password protected file. This information will be kept separate from the clinical data.

* Endoscopic Assessment: A baseline ileocolonoscopy may be additionally performed as standard of care at the discretion of the treating gastroenterologist to confirm active SBCD, either before or after the MRE. Subjects will undergo standard bowel preparation at the discretion of the treating gastroenterologist prior to ileocolonoscopy. If treatment was required after the ileocolonoscopy, treatment will not be initiated until after the baseline MRE is completed. Subjects who have had endoscopic assessment with biopsies from the ileum confirming small bowel Crohn's disease as a part of their standard of care treatment in the six (6) months prior to study enrollment may be used for the baseline study assessment, at the investigator's discretion. If a more recent endoscopic assessment is done with this reporting, the more recent assessment will be used.
* Radiological Assessment: Radiological assessment will be performed on all patients as a part of their clinical standard of care prior to initiating vedolizumab. Clinical read will be evaluated using the assessment tool in Appendix B and guidance from Appendix A.

Week 6 Visit (+/- 1 week)

Week 6 Visit assessment will be done 6 weeks (+/- 1 week) after initiating biologic as a part of clinical standard of care treatment as described in this protocol. The visit will consist of the following:

* Clinical assessment:
* Blood Tests (C-reactive, Albumin, Hematocrit, SOMAscan panel Week 14 Visit (+/- 2 weeks)

Week 14 Visit assessment will be done 14 weeks (+/- 2 weeks) after initiating biologic as a part of clinical standard of care treatment as described in this protocol. The visit will consist of the following:

* Clinical assessment:
* Physical Exam Findings: Physical exam findings will be taken from the patient's clinical care record from the most recent standard of care visit. If this data is not available from the visit, the information will be obtained from the subject during a separate visit to the clinic by the study team.
* Blood Tests (C-reactive, Albumin, Hematocrit, SOMAscan panel
* Stool Collection: As above referenced in the Baseline Visit.
* Radiological Assessment:

Phone Visit The Phone Visit assessment will be done at week 26 and 40.

- Clinical assessment: Week 52 Visit (+/- 4 weeks)

Week 52 assessments will be done 52 weeks (+/- 4 weeks) after initiating biologic as a part of clinical standard of care treatment as described in this protocol. The visit will consist of the following:

* Clinical assessment:
* Physical Exam Findings: Physical exam findings will be taken from the patient's clinical care record from the most recent standard of care visit. If this data is not available from the visit, the information will be obtained from the subject during a separate visit to the clinic by the study team.
* Blood Tests:
* Radiological Assessment: Radiological assessment will be performed on all patients as a part of their clinical standard of care. Clinical read will be evaluated using the assessment tool in Appendix B and guidance from Appendix A.
* Optional Endoscopic Assessment: Subjects can have additional endoscopic assessment as a part of their standard of care treatment, and this report may be used for the study assessment.
* Disease Progression Assessment: In order to assess the Disease Progression endpoint the following will be assessed for the time point between the Week 16 Visit MRE and the Week 52 Visit MRE:

  * Any hospitalization for disease flare or complications of the disease
  * Need for surgery related to CD
  * Need for rescue corticosteroids The treating gastroenterologists will be blinded to the results of radiological TR although they will have access to the clinical read in the electronic medical record.

ELIGIBILITY:
Inclusion:

* Patient who have had a prior standard of care (SOC) ileocolonoscopy with biopsies confirming SBCD
* And with active disease visible on a baseline MRE (small bowel only or ileocolonic disease)
* And are being initiated on a biologic (anti-TNFs, vedolizumab and ustekinumab) approved for CD, regardless of their prior biologic exposure, will be recruited.
* Prior studies have confirmed active SBCD noted on MRE as consistent with active disease using histopathology as reference standard.45

Exclusion:

* Patients who are pregnant: Subjects will not be tested for pregnancy on protocol outside of standard of care and is usually done prior to clinical radiological and endoscopic testing for patients of childbearing potential per standard of care standard operating procedures. If any subject is found to be pregnant during the study they will be discontinued from the study visit protocol and managed by primary gastroenterologist per standard of care.
* Less than 18 years of age
* Unable to provide informed consent
* Chronic kidney disease that precludes contrast administration
* Implanted medical devices that are contraindicated for MRI
* Individuals with colonic involvement without SB disease will also be excluded
* Planned surgery prior to the first follow-up MRE
* Inpatient scans will only be included if this is an MRE and adequate small bowel distension with appropriate contrast has been achieved, in the opinion of the radiology co-investigator.
* Any subject condition or situation which, in the opinion of the Investigator or regulatory authorities, interferes with optimal study participation of the participant or produces/could produce significant risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SBCD patients starting a new biologic therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Corticosteroid free remission (CFR) | 52 ± 4 weeks
  Corticosteroid free remission (CFR) will be assessed at the in-person visit at 52 ± 4 weeks where remission will be defined as using Harvey-Bradshaw index (HBI) criteria of 4 points or lower, free of any corticosteroid usage for ≥30 days.

SECONDARY OUTCOMES:
Mucosal healing (MH) | 52 ± 4 weeks.
  Secondary endpoint will be MH in the terminal ileum using criteria of Simple Endoscopic Score for Crohn's Disease (SES-CD) score of 0 to 2 at the ileocolonoscopy at 52 ± 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Parakkal Deepak, MBBS, MS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States